CLINICAL TRIAL: NCT06888284
Title: Effects of Tuijing Therapy on Heart Rate Variability and Psychological Symptoms: a Randomized Controlled Pilot Study
Brief Title: Effects of Tuijing Therapy on Heart Rate Variability and Psychological Symptoms
Acronym: TJ
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSANG Hector Wing-Hong, Chair Professor of Rehabilitation Sciences, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2024-TJ; ZH3P (Other Grant/Funding Number: the Bright Future Charitable Fund)
Record Dates: First submitted 2024-12-29; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Depression
Keywords: depression; HRV; Tui Jing
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: A pilot randomized controlled study will be conducted with Tuijing therapy as the intervention and sham therapy as the control. The intervention group will receive the actual intervention, while the sham intervention group will undergo a sham ultrasound treatment process that does not involve the active therapeutic components. A computer-generated random allocation schedule will be complied with before commencement by a person not involved in the recruitment of participants. Tuijing therapy will be administered as arm A, while the sham control group will serve as arm B. There will be a 5-day interval between interventions. Participants in arm B will receive 6 times of sham ultrasound therapy with 30 minutes each session lasting 1 month.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Screening and baseline assessments will precede the randomization process. A computerized program will generate a randomization sequence, assigning participants in a 1:1 ratio to active or sham stimulation. To ensure concealment, opaque sealed envelopes will be used, managed by a research assistant not involved in the direct handling of the study. While it is impossible to blind the therapist due to the intervention's nature, assessors will remain unaware of the treatment assignments. To evaluate the effectiveness of the blinding, participants and assessors will be asked two questions at the study's conclusion: "What type of treatment do you believe you/the participant received?" and "How confident are you that you received active stimulation?" The latter will be rated on a scale from 0 (no confidence) to 10 (very confident), aiming to measure their perceptions and confidence regarding the treatment received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- The Tui Jing Group (Experimental): Tui Jing group:
  A standardized treatment protocol targeting specific meridians identified in traditional Chinese medicine will be followed. Designed specifically for psychological symptoms, the protocol involves bilateral therapy on four key meridians. These include the Hand Shaoyin Heart Meridian, Hand Jueyin Pericardium Meridian, Foot Taiyin Spleen Meridian, and Foot Jueyin Liver Meridian.
  Interventions: Behavioral: Tui Jing therapy
- The Sham control (Sham Comparator): Participants will receive a sham ultrasound intervention on the same meridians. To enhance comfort and prevent cold sensations from the metal probe, the ultrasound device will be pre-warmed to body temperature. A gel, mimicking the texture of the lubricant used in Tui Jing therapy, will be applied. The device will mimic the motion, direction, duration, and frequency of the Tui Jing therapy, but without activating the ultrasound's therapeutic mode. The participants will be informed that they are accepting low-intensity ultrasound mode, which will not produce any sensory perception, ensuring they can't distinguish between the active and the sham interventions.
  Interventions: Device: sham ultrasound intervention

INTERVENTIONS:
Behavioral: Tui Jing therapy — Tui Jing therapy (Gua Sha + Meridian pressure) was utilized, a specialized form of Gua Sha that incorporates traditional techniques with targeted pressure on specific meridians.
  Arms: The Tui Jing Group
Device: sham ultrasound intervention — Participants will receive a sham ultrasound intervention on the same meridians. To enhance comfort and prevent cold sensations from the metal probe, the ultrasound device will be pre-warmed to body temperature. A gel, mimicking the texture of the lubricant used in Tui Jing therapy, will be applied. The device will mimic the motion, direction, duration, and frequency of the Tui Jing therapy, but without activating the ultrasound's therapeutic mode. The participants will be informed that they are accepting low-intensity ultrasound mode, which will not produce any sensory perception, ensuring in distinguishing ability between active and sham interventions
  Arms: The Sham control

SUMMARY:
Background Mental disorders are recognized as a major cause of disability and disease burden across the lifespan. Gua Sha is believed to improve mental health and sleep quality significantly. Tui Jing is an innovative type of Gua Sha therapy that penetrates deep into the muscles and fascia rather than just acting on the surface of the skin. Modern research has revealed that Gua Sha is extensively utilized for pain-related symptoms, and its therapeutic effects may be attributed to anti-inflammatory and immunomodulatory mechanisms. Although Gua Sha has demonstrated efficacy in treating various diseases, limited research exists regarding its impact and underlying mechanisms on mental health. This study will conduct a pilot clinical trial to assess the efficacy of Tuijing Therapy on mental health. Autonomic function is closely associated with psychological symptoms, and HRV reflects the activation of the vagus nerve. This study aims to obtain preliminary evidence that Gua Sha can modulate HRV by regulating vagal function, potentially ameliorating psychological disorders.

Population A formal sample size estimation is not required for pilot feasibility studies because the primary objective of this study is to assess feasibility and acceptance. The sample size is estimated according to a method for preliminary pilot study. The researchers aim to recruit 36 participants to assess the feasibility of the study. Adults without any chronic diseases who score over 14 on the HAM-D 17 and have no smoking or drinking habits will be included.

Method A pilot randomized controlled study will be conducted with Tuijing therapy as the intervention and sham therapy as the control. The intervention group will receive the actual intervention, while the sham intervention group will undergo a sham ultrasound treatment process that does not involve the active therapeutic components. A computer-generated random allocation schedule will be complied with before commencement by a researcher not involved in recruiting participants. Tuijing therapy will be administered as arm A, while the sham control group will serve as arm B. There will be a 5-day interval between interventions. Participants in arm B will receive 6 times of sham ultrasound therapy with 30 minutes each session lasting 1 month. Participants in arm A will receive 6 times of Tui Jing therapy with 30 minutes each session lasting 1 month. Heart rate variability, brain activity, skin reflection, pain perception, psychological symptoms, and sleep quality will be assessed as outcome measures.

Outcomes The primary outcomes of this study are feasibility, acceptance, and satisfaction. As secondary outcomes, this study will assess changes in heart rate variability, brain activity, skin reflection, pain perception, psychological symptoms, and sleep quality. Heart rate variability will be measured using a heart rate variability monitoring device, sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), and psychological symptoms will be evaluated using several related scales.

DETAILED DESCRIPTION:
Procedures The researcher will conduct an initial telephone interview to provide study information and screen potential participants for eligibility. Each participant will receive full details about the study's purpose and will be required to sign an informed consent form. All participants will be invited for two in-person sessions before accepting any intervention. In the first session, comprehensive medical histories, brief semi-structured interviews for psychological symptoms, clinical examinations, general information, and questionnaires will be conducted to determine eligibility. Eligible participants in the first session will be included in the second session. The second session will be scheduled to collect baseline data for further analysis. Eligible participants meeting inclusion criteria will be randomly assigned to receive either Tui Jing therapy or sham stimulation. The intervention will be conducted by a qualified therapist (with a qualification in TCM [Master's and Bachelor's degree in Traditional Chinese medicine]) from the Department of Rehabilitation Sciences at PolyU, while another qualified researcher will be responsible for clinical interviews, screening, and data collection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 55 years old
* Willingness to participate in the study and undergo randomization
* Proficiency in Chinese
* Absence of severe chronic diseases
* Experience with depression symptoms for over three months
* Scoring 20 or higher on the Montreal Cognitive Assessment (MoCA)
* Scoring above 14 on the Hamilton Depression Rating Scale 17

Exclusion Criteria:

* The presence of cardiovascular disease (CVD)
* Severe head trauma, intracranial hypertension, implanted ferromagnetic devices, or a history of epilepsy
* Engagement in any pharmacological or non-pharmacological treatments within the past month
* Existing skin conditions or susceptibility to skin injuries
* Any form of cognitive impairment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Satisfaction | through study completion, an average of 6 months
  Treatment Satisfaction Score
  Measurement: 10-point numerical rating scale (0 = "Completely Dissatisfied", 10 = "Fully Satisfied") Unit: Scale score (0-10) Tool: Standardized questionnaire
Intervention Liking Rate | through study completion, an average of 6 months
  Intervention Liking Rate
  Measurement: Binary response (Yes/No) Unit: Percentage (% "Yes" responses) Tool: Structured interview
Recommendation Willingness Rate | through study completion, an average of 6 months
  Recommendation Willingness Rate
  Measurement: Binary response (Yes/No) Unit: Percentage (% "Yes" responses) Tool: Structured interview
Eligibility Rate | through study completion, an average of 6 months
  Eligibility Rate
  Formula: (Number of eligible individuals / Total screened) × 100% Unit: Percentage (%) Data Source: Screening records
Recruitment Rate | through study completion, an average of 6 months
  Recruitment Rate
  Formula: (Number of consented participants / Eligible individuals) × 100% Unit: Percentage (%) Data Source: Recruitment database
Retention Rate | through study completion, an average of 6 months
  Retention Rate
  Formula: (Number of completers / Enrolled participants) × 100% Unit: Percentage (%) Data Source: Follow-up records
Adverse Event Rate | through study completion, an average of 6 months
  Adverse Event Rate
  Formula: (Participants reporting adverse events / Total participants) × 100% Unit: Percentage (%) Data Source: Adverse event report forms
Attrition Rate | through study completion, an average of 6 months
  Attrition Rate
  Formula: (Number of withdrawals / Enrolled participants) × 100% Unit: Percentage (%) Data Source: Withdrawal documentation
Adherence Rate | through study completion, an average of 6 months
  Adherence Rate
  Formula: (Days of full protocol adherence / Total intervention days) × 100% Unit: Percentage (%) Data Source: Intervention logs

SECONDARY OUTCOMES:
Psychological outcomes - Depression symptoms | through study completion, an average of 6 months
  Hamilton Depression Rating Scale (HAMD-17)
  Scale Range: 0-52 points Interpretation: Higher scores indicate greater depression severity Assessment: Semi-structured interview by trained raters Time Frame: Baseline, monthly during intervention, post-intervention
Psychological outcomes - Depression symptoms | through study completion, an average of 6 months
  Patient Health Questionnaire (PHQ-9)
  Scale Range: 0-27 points Interpretation: Higher scores indicate greater depression severity Assessment: Self-administered questionnaire
Sleep quality | From date of randomization until two weeks after the last treatment
  Pittsburgh Sleep Quality Index (PSQI)
  Scale Range: 0-21 points Interpretation: Higher scores indicate poorer sleep quality Assessment: Standardized self-report questionnaire
Sleep Efficiency | From date of randomization until two weeks after the last treatment
  Objective Sleep Efficiency
  Measurement: (Total sleep time / Time in bed) × 100% Unit: Percentage (%) Tool: Fitbit Inspire 2 (FDA-cleared wearable device) Data Collection: Automated daily sync to the research platform
Subjective Sleep Quality | From date of randomization until two weeks after the last treatment
  Measurement: 10-point Likert scale (1 = "Very Poor", 10 = "Excellent") Unit: Scale score (1-10) Tool: Standardized sleep diary
Heart Rate Variability (HRV) | through study completion, an average of 6 months
  Metrics:
  RMSSD (Root Mean Square of Successive Differences) SDNN (Standard Deviation of NN Intervals) Low Frequency (LF: 0.04-0.15 Hz) High Frequency (HF: 0.15-0.40 Hz)
  Unit: Milliseconds (ms) Tool: NeXus-10 Biofeedback System (Mind Media) Protocol: 10-minute resting-state measurement
Skin Reactions | through study completion, an average of 6 months
  Skin Discoloration Severity
  Measurement Protocol:
  Capture multispectral images using the IBOOLO DE-4100 system Calculate the ΔContrast between affected and normal skin areas Formula: ΔContrast = |Mean lesion chroma value - Mean normal skin chroma value| Unit: Standardized chroma difference (0-100; 0=no difference, 100=maximal difference)
  Quality Control:
  Imaging environment: Standardized D65 lighting Analysis software: IBOOLO SkinAnalyzer Pro v3.2

CONTACTS AND LOCATIONS:
Locations (1):
- Polyu, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Confidentiality Agreement